CLINICAL TRIAL: NCT05049473
Title: Treatment of Mature B-ALL and Burkitt Lymphoma (BL) in Adult Patients. BURKIMAB-14.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Collaborators: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BURKIMAB-14
Record Dates: First submitted 2021-09-08; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Mature B-Cell Leukemia Burkitt Type; Burkitt Lymphoma (BL); Unclassifiable Lymphoma Between DCBL and BL
Keywords: Mature B-ALL; Burkitt lymphoma; Adult
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Rituximab; Methotrexate; Dexamethasone; Ifosfamide; Vincristine; Etoposide; Cytarabine; Cyclophosphamide; Doxorubicin; Vindesine; Hydrocortisone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Pts with biological age up to 55 y with advanced stage will receive 6 cycles of intensive treatment: blocks (A1-B1-C1-A2-B2-C2). If after A1 and B1 cycles CR is observed, the rest of the cycles will be administered with reduced doses.
  In pts with biological age >55 y with advanced stage block will receive A and B with attenuated doses (A1*-B1*-A2*-B2*-A3*-B3*).
  Pts with biological age up to 55 y with localized stage (non-bulky I or II) with CR after 2 cycles will finish treatment after 4 blocks. If CR is not reached, patients will complete the 6 treatment cycles.
  Pts with a biological age >55 y with localized stage (non-bulky I or II) with CR after 2 cycles will finish treatment after 4 attenuated blocks (A1*-B1*-A2*-B2*). If CR is not reached, patients will complete the 6 cycles of treatment.
  Interventions: Drug: Rituximab; Drug: Methotrexate; Drug: Dexamethasone; Drug: Iphosphamid; Drug: Vincristine; Drug: Etoposide; Drug: Cytarabine; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vindesine; Drug: Hydrocortisone; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m² IV. Day 1. Cycles: A1/A1*, B1/B1*, C1/A2*, A2/B2*, B2/A3*, C2/B3*. Two additional doses after 6 cycles in case of localized stage patients without CR after four cycles or advanced stage patients.
Drug: Methotrexate — Methotrexate 1500 mg/m² IV 24h-infusion. Day 2. Cycles: A1, B1, C1 (1000 mg/m² if patient in CR) , A2 (1000 mg/m² if patient in CR), B2 (1000 mg/m² if patient in CR) , C2 (1000 mg/m² if patient in CR) Methotrexate 500 mg/m² IV 24h-infusion. Day 2. Cycles: A1*, B1*, A2*, B2*, A3*, B3*
Drug: Dexamethasone — Dexamethasone 10 mg/m² PO or IV bolus. Days: 2 to 6. Cycles: A1/A1*, B1/B1*, C1/A2*, A2/B2*, B2/A3*, C2/B3*.
Drug: Iphosphamid — Iphosphamid 800 mg/m² IV in 1 hour. Days: 2 to 6. Cycles: A1, A2 (500 mg/m² if patient in CR).
  Iphosphamid 400 mg/m² IV in 1 hour. Days: 2 to 6. Cycles: A1*.
Drug: Vincristine — Vincristine 2 mg IV bolus. Day 2. Cycles: A1, B1, A2, B2 Vincristine 1 mg IV bolus. Day 2. Cycles: B1*, B2*, B3*
Drug: Etoposide — Etoposide (VP16) 100 mg/m² IV in 1 hour. Days: 5, 6. Cycle: A1, A2. Etoposide (VP16) 250 mg/m² IV in 1 hour. Days: 5, 6. Cycle: C1, C2. Etoposide (VP16) 60 mg/m² IV in 1 hour. Days: 5, 6. Cycle: A1*, A2*, A3*.
Drug: Cytarabine — Cytarabine 150 mg/m² IV in 1 hour every 12 hours. Days: 5, 6. Cycles: A1, A2 Cytarabine 2 g/m² IV in 3 hours every 12 hours. Day: 6. Cycle: C1 (1.5 g/m² if patient in CR), C2 (1.5 g/m² if patient in CR) Cytarabine 60 mg/m² IV in 1 hour every 12 hours. Days: 5, 6. Cycles: A1*, A2*, A3*
Drug: Cyclophosphamide — Cyclophosphamide 200 mg/m² IV in 1 hour. Days 1 to 5. Pre-phase. Cyclophosphamide 200 mg/m² IV in 1 hour. Days 2 to 6. Cycles: B1, B2, B1*, B2*, B3*
Drug: Doxorubicin — Doxorubicin 25 mg/m² IV in 15 min. Days 5 and 6. Cycles: B1/B1*, B2, B2*, B3*
Drug: Vindesine — Vindesine 3 mg/m2 (max 5 mg) IV bolus. Day 2. Cycles: C1, C2
Drug: Cytarabine — Cytarabine 30 mg IT. Days 2 and 6. Cycles A1, B1, A2, B2
Drug: Methotrexate — Methotrexate 12 mg IT. Day 1. Pre-phase Methotrexate 12 mg IT. Days 2 and 6. Cycles: A1, B1, A2, B2 Methotrexate 15 mg IT. Day 2. Cycles: A1*, B1*, A2*, B2*, A3*, B3*
Drug: Hydrocortisone — Hydrocortisone 20 mg IT. Days 2 and 6. Cycles: A1, B1, A2, B2
Drug: Prednisone — Prednisone 60 mg/m2 PO or IV bolus. Days 1 to 5. Pre-phase.

SUMMARY:
Rituximab combined with a specific intensive chemotherapy is considered the standard treatment for newly diagnosed patients with mature B leukemia/lymphoma. However, the toxicity of this therapy is high. The purpose of this trial is to reduce the dose intensity of the chemotherapy blocks once the patient has achieved complete response. With this approach the investigators expect to maintain the efficacy and to reduce the toxicity of the chemotherapy, specially the rate of deaths in complete response.

DETAILED DESCRIPTION:
Patients younger than 55 years in complete response after two blocks of rituximab and specific intensive chemotherapy will receive four additional blocks of rituximab and attenuated chemotherapy (reduction by 33% of the dose of cyclophosphamide, methotrexate and cytarabine) followed by additional rituximab doses as consolidation. Patients older than 55 years will receive the six blocks with attenuated chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients diagnosed with de novo mature B-ALL, Burkitt lymphoma (BL). Under physician's criteria, patients with unclassified B-lymphoma with intermediate characteristics between DLBCL and BL could be included.
* Candidate to intensive treatment.

Exclusion Criteria:

* Other ALL subtype different from mature B-ALL/BL
* Severe complications not due to mature B-ALL/BL (eg, sepsis, pneumonia, shock or hemorrhage) at diagnosis.
* Renal failure not due to mature B-ALL /BL
* Heart or liver failure
* Severe lung disease
* Secondary mature B-ALL/BL
* Hypersensitivity to foreign proteins
* Previous treatment with cytotoxic drugs
* Pregnancy/breastfeeding
* Severe psychiatric disease
* Lack of social or familiar support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Throughout the study period. Approximately 3 years
  Defined as the time from diagnosis to death by any cause or last follow-up.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Throughout the study period. Approximately 3 years
  Defined as the time from diagnosis to progression disease, relapse or death by any cause or last follow-up.
Number of patients with toxicity during the treatment period. | Throughout the study period. Approximately 3 years
  Number of patients experiencing different toxicities during the treatment period, classified according to severity and graded according to NCTCAE V4.0

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP MARIA RIBERA SANTASUSANA, M.D.; Ph.D., Study Chair — ICO-Hospital Germans Trias i Pujol; JUAN MANUEL SANCHO CIA, M.D.; Ph.D., Study Chair — ICO-Hospital Germans Trias i Pujol
Locations (29):
- Spain (29):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO-Hospital Duran i Reynals, Bellvitge
  - Hospital Universitario de Basurto, Bilbao
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Universitario de Gran Canaria Dr Negrín, Las Palmas de Gran Canaria
  - Hospital Arnau de Vilanova (Lleida), Lleida
  - Hospital 12 De Octubre, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital La Zarzuela, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Clínico de Málaga, Málaga
  - Hospital Central de Asturias, Oviedo
  - Son Llàtzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - Complexo Hospitalario Santiago de Compostela, Santiago de Compostela
  - ICO-Hospital Joan XXIII, Tarragona
  - Mútua de Terrassa, Terrassa
  - Hospital Universitario de Torrejón, Torrejón de Ardoz
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Background] Sancho JM, Ribera JM. Linfoma de Burkitt. En: Manual Práctico de Hematología Clínica. 4ª edición 2012.
- [Background] WHO Classification of Tumours of Haematopoietics and Lymphoid Tissues, 2008.
- [Background] Karantanis D, Durski JM, Lowe VJ, Nathan MA, Mullan BP, Georgiou E, Johnston PB, Wiseman GA. 18F-FDG PET and PET/CT in Burkitt's lymphoma. Eur J Radiol. 2010 Jul;75(1):e68-73. doi: 10.1016/j.ejrad.2009.07.035. Epub 2009 Aug 27. PMID 19716248
- [Background] Zeng W, Lechowicz MJ, Winton E, Cho SM, Galt JR, Halkar R. Spectrum of FDG PET/CT findings in Burkitt lymphoma. Clin Nucl Med. 2009 Jun;34(6):355-8. doi: 10.1097/RLU.0b013e3181a34552. PMID 19487844
- [Background] Just PA, Fieschi C, Baillet G, Galicier L, Oksenhendler E, Moretti JL. 18F-fluorodeoxyglucose positron emission tomography/computed tomography in AIDS-related Burkitt lymphoma. AIDS Patient Care STDS. 2008 Sep;22(9):695-700. doi: 10.1089/apc.2008.0174. PMID 18793085
- [Background] Hoelzer D, Ludwig WD, Thiel E, Gassmann W, Loffler H, Fonatsch C, Rieder H, Heil G, Heinze B, Arnold R, Hossfeld D, Buchner T, Koch P, Freund M, Hiddemann W, Maschmeyer G, Heyll A, Aul C, Faak T, Kuse R, Ittel TH, Gramatzki M, Diedrich H, Kolbe K, Fuhr HG, Fischer K, Schadeck-Gressel C, Weiss A, Strohscheer I, Metzner B, Fabry U, Gokbuget N, Volkers B, Messerer D, Uberla K. Improved outcome in adult B-cell acute lymphoblastic leukemia. Blood. 1996 Jan 15;87(2):495-508. PMID 8555471
- [Background] Reiter A, Schrappe M, Tiemann M, Ludwig WD, Yakisan E, Zimmermann M, Mann G, Chott A, Ebell W, Klingebiel T, Graf N, Kremens B, Muller-Weihrich S, Pluss HJ, Zintl F, Henze G, Riehm H. Improved treatment results in childhood B-cell neoplasms with tailored intensification of therapy: A report of the Berlin-Frankfurt-Munster Group Trial NHL-BFM 90. Blood. 1999 Nov 15;94(10):3294-306. PMID 10552938
- [Background] Thomas DA, Cortes J, O'Brien S, Pierce S, Faderl S, Albitar M, Hagemeister FB, Cabanillas FF, Murphy S, Keating MJ, Kantarjian H. Hyper-CVAD program in Burkitt's-type adult acute lymphoblastic leukemia. J Clin Oncol. 1999 Aug;17(8):2461-70. doi: 10.1200/JCO.1999.17.8.2461. PMID 10561310
- [Background] Adde M, Shad A, Venzon D, Arndt C, Gootenberg J, Neely J, Nieder M, Owen W, Seibel N, Wilson W, Horak ID, Magrath I. Additional chemotherapy agents improve treatment outcome for children and adults with advanced B-cell lymphomas. Semin Oncol. 1998 Apr;25(2 Suppl 4):33-9; discussion 45-8. PMID 9578060
- [Background] Lee EJ, Petroni GR, Schiffer CA, Freter CE, Johnson JL, Barcos M, Frizzera G, Bloomfield CD, Peterson BA. Brief-duration high-intensity chemotherapy for patients with small noncleaved-cell lymphoma or FAB L3 acute lymphocytic leukemia: results of cancer and leukemia group B study 9251. J Clin Oncol. 2001 Oct 15;19(20):4014-22. doi: 10.1200/JCO.2001.19.20.4014. PMID 11600602
- [Background] Ribera JM, Garcia O, Grande C, Esteve J, Oriol A, Bergua J, Gonzalez-Campos J, Vall-Llovera F, Tormo M, Hernandez-Rivas JM, Garcia D, Brunet S, Alonso N, Barba P, Miralles P, Llorente A, Montesinos P, Moreno MJ, Hernandez-Rivas JA, Bernal T. Dose-intensive chemotherapy including rituximab in Burkitt's leukemia or lymphoma regardless of human immunodeficiency virus infection status: final results of a phase 2 study (Burkimab). Cancer. 2013 May 1;119(9):1660-8. doi: 10.1002/cncr.27918. Epub 2013 Jan 29. PMID 23361927
- [Background] Hoelzer D, Walewski J, Döhner H, Schmid M, Hiddemann W, Baumann A, et al. Substantially improved outcome of adult Burkitt Non-Hodgkin lymphoma and leukemia patients with rituximab and a short-intensive chemotherapy; Report of a large prospective multicenter trial. Fifty-four annual meeting of American Society of Hematology. Abstract 667
- [Background] Intermesoli T, Rambaldi A, Rossi G, Delaini F, Romani C, Pogliani EM, Pagani C, Angelucci E, Terruzzi E, Levis A, Cassibba V, Mattei D, Gianfaldoni G, Scattolin AM, Di Bona E, Oldani E, Parolini M, Gokbuget N, Bassan R. High cure rates in Burkitt lymphoma and leukemia: a Northern Italy Leukemia Group study of the German short intensive rituximab-chemotherapy program. Haematologica. 2013 Nov;98(11):1718-25. doi: 10.3324/haematol.2013.086827. Epub 2013 Jun 10. PMID 23753030
- [Background] Oriol A, Ribera JM, Esteve J, Sanz MA, Brunet S, Garcia-Boyero R, Fernandez-Abellan P, Marti JM, Abella E, Sanchez-Delgado M, Penarrubia MJ, Besalduch J, Moreno MJ, Borrego D, Feliu E, Ortega JJ; PETHEMA Group, Spanish Society of Hematology. Lack of influence of human immunodeficiency virus infection status in the response to therapy and survival of adult patients with mature B-cell lymphoma or leukemia. Results of the PETHEMA-LAL3/97 study. Haematologica. 2003 Apr;88(4):445-53. PMID 12681972
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Bleyer WA. New vistas for leucovorin in cancer chemotherapy. Cancer. 1989 Mar 15;63(6 Suppl):995-1007. doi: 10.1002/1097-0142(19890315)63:6+3.0.co;2-r. PMID 2645044
- [Background] Pauley JL, Panetta JC, Crews KR, Pei D, Cheng C, McCormick J, Howard SC, Sandlund JT, Jeha S, Ribeiro R, Rubnitz J, Pui CH, Evans WE, Relling MV. Between-course targeting of methotrexate exposure using pharmacokinetically guided dosage adjustments. Cancer Chemother Pharmacol. 2013 Aug;72(2):369-78. doi: 10.1007/s00280-013-2206-x. Epub 2013 Jun 13. PMID 23760811
- [Background] Reiter A, Schrappe M, Ludwig WD, Tiemann M, Parwaresch R, Zimmermann M, Schirg E, Henze G, Schellong G, Gadner H, Riehm H. Intensive ALL-type therapy without local radiotherapy provides a 90% event-free survival for children with T-cell lymphoblastic lymphoma: a BFM group report. Blood. 2000 Jan 15;95(2):416-21. PMID 10627444
- [Background] Pauley JL, Panetta JC, Schmidt J, Kornegay N, Relling MV, Pui CH. Late-onset delayed excretion of methotrexate. Cancer Chemother Pharmacol. 2004 Aug;54(2):146-52. doi: 10.1007/s00280-004-0797-y. Epub 2004 May 18. PMID 15148625
- [Background] Pinedo HM, Zaharko DS, Bull JM, Chabner BA. The reversal of methotrexate cytotoxicity to mouse bone marrow cells by leucovorin and nucleosides. Cancer Res. 1976 Dec;36(12):4418-24. PMID 1087180
- [Background] Scott JR, Zhou Y, Cheng C, Ward DA, Swanson HD, Molinelli AR, Stewart CF, Navid F, Jeha S, Relling MV, Crews KR. Comparable efficacy with varying dosages of glucarpidase in pediatric oncology patients. Pediatr Blood Cancer. 2015 Sep;62(9):1518-22. doi: 10.1002/pbc.25395. Epub 2015 Jan 28. PMID 25631103
- [Derived] Ribera JM, Morgades M, Garcia-Calduch O, Sirvent M, Buendia B, Cervera M, Luzardo H, Hernandez-Rivas JM, Sitges M, Garcia-Cadenas I, Abrisqueta P, Montesinos P, Bastos-Oreiro M, De Llano MQ, Bravo P, Torrent A, Herrera P, Garcia-Guinon A, Vall-Llovera F, Serrano J, Terol MJ, Bergua JM, Garcia-Noblejas A, Barrenetxea C, Llorente L, Garcia-Belmonte D, Gimeno E, Cladera A, Mercadal S, Sancho JM. Feasibility and outcomes after dose reduction of immunochemotherapy in young adults with Burkitt lymphoma and leukemia: results of the BURKIMAB14 trial. Haematologica. 2024 Feb 1;109(2):543-552. doi: 10.3324/haematol.2023.283342. PMID 37560813